CLINICAL TRIAL: NCT03366727
Title: Drug-eluting Balloon for Arteriovenous Fistula in China
Brief Title: AcoArt III / Arterio-venous Fistula in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acotec-05
Record Dates: First submitted 2017-10-27; First posted 2017-12-08 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Arteriovenous Fistula Stenosis
Keywords: drug eluting balloon

STUDY DESIGN:
Intervention Model Description: one arm treated with drug-coated balloon catheter, the other arm treated with plain balloon catheter
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB group (Experimental): this group treated with drug coated balloon catheter, Orchid
  Interventions: Device: drug-coated balloon catheter （Orchid, Acotec）
- PTA group (Experimental): this group treated with plain balloon catheter, Admiral Xtreme
  Interventions: Device: plain balloon catheter (Admiral, medtronic)

INTERVENTIONS:
Device: drug-coated balloon catheter （Orchid, Acotec） — After predilation, using drug-coated balloon catheter to cover the whole treated segment
  Arms: DCB group
Device: plain balloon catheter (Admiral, medtronic) — After predilation, using plain balloon catheter to cover the whole treated segment
  Arms: PTA group

SUMMARY:
This trial is aimed to evaluate the safety and efficacy of DCB in treating AVF stenosis in chinese population.

DETAILED DESCRIPTION:
For years, first-line treatment of AVFs stenoses has been percutaneous transluminal angioplasty. However, restenosis and reintervention rates remain incredibly high and occur, according to recent studies, in up to 60% and 70% of patients at 6 and 12 months, respectively. Drug-coated balloons delivering paclitaxel at the angioplasty site have proved their superiority in the treatment of coronary and peripheral arterial stenoses. Paclitaxel reduces neointimal hyperplasia and drug-coated balloons,therefore, it represents an attractive option for AVF stenoses.

ELIGIBILITY:
Inclusion Criteria:

* Age during 18-85 years old
* Arteriovenous fistula is matured and has undergone one or more hemodialysis sessions
* Venous stenosis of the AV fistula
* target lesion has stenosis ≥50% evidenced by angiography. and have at least one symptom of these：1,the venous pressure increased significantly during dialysis. 2,abnormal physical examination. 3,Decrease in blood flow
* the length of target lesion ≤100mm
* Patient able to give informed consent
* residual stenosis ≤30% after predilation

Exclusion Criteria:

* Women who are breastfeeding, pregnant or are intending to become pregnant
* AVF located at lower limbs
* two or more than two stenosis at the target vessel.
* Obstruction of central venous return
* ISR
* AVF with acute thrombosis requiring lysis or thrombectomy in 30 days
* vascular access has surgery in 30 days or intending to undergo a surgery
* known hypersensitivity to aspirin, heparin, clopidogrel,paclitaxel, contrast medium, etc.
* Patients undergoing immunotherapy or suspected / confirmed vasculitis
* Patients with history of blood coagulation dysfunction and history of thrombocytopenic purpura
* Vascular access infection or systemic active infection
* patients's life expectancy is less than 12 months
* Renal transplantation has been planned or converted to peritoneal dialysis
* Other medical conditions that lead to researchers who believe that patients may not be able to follow the trial program
* involved in other drugs, biology, medical device research, or has been involved in other similar products clinical Test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
primary patency of target lesion in 6 months | 6 months
  Primary Patency is defined as the freedom of reintervention for the target lesion,including: 1)clinical driven target lesion reintervention;2)thrombus formation in target lesion; 3) surgical removal of target lesion;4) AVF was abandoned because of the target lesion could not be retreated

SECONDARY OUTCOMES:
primary patency of target lesion in 12 months | 12 months
  Primary Patency is defined as the freedom of reintervention for the target lesion,including: 1)clinical driven target lesion reintervention;2)thrombus formation in target lesion; 3) surgical removal of target lesion;4) AVF was abandoned because of the target lesion could not be retreated
number of reinterventions | 12 months
  number of reinterventions in 12 months
device success | during the procedure
  Successful delivery to the target lesion, deployment, and retrieval at index procedure
clinical success | 5 days
  The resumption of dialysis for at least one session after the index procedure
Procedural Success | 2 weeks
  residual stenosis≤30% and absence of SAE during perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Principal Investigator — Chinese PLA General Hospital; Lan Zhang, Principal Investigator — RenJi Hospital
Locations (13):
- China (13):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Tongren hospital, Capital medical university, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong provincial people's hospital, Guangzhou, Guangdong
  - Nanfang hospital, Guangzhou, Guangzhou
  - The first hospital of Hebei medical university, Shijiangzhuang, Hebei
  - The first hospital of Chinese medical university, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The first hospital of Jilin medical university, Changchun, Jilin
  - Renji Hospital ShangHai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - Shaoyifu hospital, zhejiang medical universiyt, Hangzhou, Zhejiang
  - Zhejiang provincial people's hospital, Hangzhou, Zhejiang
  - Beijing Friendship Hospital,Capital Medical University, Beijing

REFERENCES:
- [Derived] Zhao Y, Wang P, Wang Y, Zhang L, Zhao Y, Li H, He Q, Liu H, Luo J, Jia X, Yu Z, Guo W, Zhang L. Drug-Coated Balloon Angioplasty for Dysfunctional Arteriovenous Hemodialysis Fistulae: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2024 Mar 1;19(3):336-344. doi: 10.2215/CJN.0000000000000359. Epub 2023 Dec 18. PMID 38191561